CLINICAL TRIAL: NCT04764448
Title: A Phase 2, Randomized, Double-blind, Placebo-Controlled Study Investigating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Two Dose Levels of Belcesiran in Patients With Alpha-1 Antitrypsin Deficiency-Associated Liver Disease
Brief Title: A Study of Belcesiran in Patients With AATLD
Acronym: ESTRELLA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Development project was discontinued
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DCR-A1AT-201
Record Dates: First submitted 2021-01-27; First posted 2021-02-21 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Belcesiran Cohort 1 (Experimental)
  Interventions: Drug: Belcesiran
- Placebo Cohort 1 (Placebo Comparator)
  Interventions: Other: Placebo
- Belcesiran Cohort 2 (Experimental)
  Interventions: Drug: Belcesiran
- Placebo Cohort 2 (Placebo Comparator)
  Interventions: Other: Placebo
- Belcesiran Cohort 3 (Experimental)
  Interventions: Drug: Belcesiran
- Placebo Cohort 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Belcesiran — Administered multiple fixed doses of belcesiran by subcutaneous (sc) injection for 24 weeks. Extension offered to participants.
  Arms: Belcesiran Cohort 1
Other: Placebo — Comparator: Placebo Cohort 1 Administered sterile normal saline (0.9% NaCl) matching volume of belcesiran by subcutaneous (sc) injection for 24 weeks. Extension offered to participants.
  Arms: Placebo Cohort 1
Drug: Belcesiran — Administered multiple fixed doses of belcesiran by subcutaneous (sc) injection for 48 weeks. Extension offered to participants.
  Arms: Belcesiran Cohort 2
Other: Placebo — Administered sterile normal saline (0.9% NaCl) matching volumes of belcesiran by subcutaneous (sc) injection for 48 weeks. Extension offered to participants.
  Arms: Placebo Cohort 2
Drug: Belcesiran — Administered multiple fixed doses of belcesiran by subcutaneous (sc) injection for 96 weeks.
  Arms: Belcesiran Cohort 3
Other: Placebo — Administered sterile normal saline (0.9% NaCl) matching volumes of belcesiran by subcutaneous (sc) injection for 96 weeks.
  Arms: Placebo Cohort 3

SUMMARY:
This is a multiple dose, randomized, placebo-controlled, double-blind study of belcesiran to evaluate the safety, tolerability, PK, and PD in adult patients with PiZZ AATD-associated liver disease (AATLD).

The study will be conducted in 3 separate cohorts. A total of up to 16 participants may be enrolled in Cohort 1 and 2. A total number of 30 subjects will be enrolled in cohort 3. The 3 cohorts are differentiated by the duration of the treatment period, the number of doses administered, and the timing of the second liver biopsy.

DETAILED DESCRIPTION:
AATD-associated liver disease is a progressive condition resulting in liver fibrosis, cirrhosis, and in some cases hepatocellular carcinoma. The lack of functional alpha-1 antitrypsin (AAT) in individuals with the PiZZ genotype, in conjunction with other precipitating factors, can lead to unchecked activity of neutrophil elastases in the alveoli; causing emphysema and chronic obstructive pulmonary disease (COPD). This loss-of-function mechanism may be addressed by use of intravenous augmentation therapy, which aims to substitute the missing AAT by infusing alpha-1 proteinase inhibitor (A1PI), purified from pooled human plasma.

While augmentation therapy can address the loss of AAT in the lung, no treatment exists for the associated liver disease.

Given the severity of the disease, with approximately 10% of affected patients developing liver cirrhosis and a subgroup of those patients in need of liver transplantation, and the lack of an effective treatment that addresses the toxic hepatic "gain-of-function" mechanism, there is an urgent unmet medical need to develop a therapy that can help this particular patient population.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years, inclusive, at the time of consent.
* Documented diagnosis of PiZZ-type alpha-1 antitrypsin deficiency, confirmed by genotyping. Historical genotyping data may be used, if available.
* AATD-associated liver disease documented by liver biopsy at Screening.
* Consent to undergo paired liver biopsies.
* Lung, renal and liver function within acceptable limits
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* History of chronic liver disease other than non-alcoholic fatty liver disease from any cause other than PiZZ-type alpha-1 antitrypsin deficiency.
* Child-Pugh Score B or C.
* History of one single severe exacerbation of underlying lung disease in the year prior to randomization.
* History of clinically significant respiratory infections (including pneumonia and lower respiratory tract infections), as determined by the Investigator, in the 3 months prior to screening
* Use of an RNAi drug at any time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2024-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bowman, MD, Study Director — Dicerna Pharmaceuticals / Novo Nordisk
Locations (23):
- United States (3):
  - University of California - San Diego, La Jolla, California
  - University of Florida, Gainesville, Florida
  - Medical University of South Carolina, Charleston, South Carolina
- St Vincent's Hospital Melbourne, Melbourne, Australia
- Medizinische Universitaet Innsbruck, Innsbruck, Austria
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec, Canada
- CHU Bordeaux - Hopital Haut-Leveque - Centre François Magendie, Pessac, France
- Germany (2):
  - Universitaetsklinikum Aachen, AoeR, Aachen
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
- Beaumont Hospital, Dublin, Ireland
- Leiden University Medical Center, Leiden, Netherlands
- New Zealand (2):
  - Auckland Clinical Studies, Grafton, Auckland
  - Waikato Hospital, Hamilton
- Portugal (3):
  - Hospital da Senhora da Oliveira - Guimaraes, Creixomil
  - Centro Hospitalar Universitario de Sao Joao, Porto
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, EPE, Vila Real
- Spain (2):
  - Hospital Universitario Marques de Valdecilla Santander, Santander, Cantabria
  - Hospital Universitario La Paz, Madrid
- CTC Clinical Trial Consultants AB Uppsala, Uppsala, Sweden
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge University, Cambridge
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Free London NHS Foundation Trust, Royal Free Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 8 sites in 8 countries. The number of sites that randomised participants are as follows: Australia (1), Belgium (1), Germany (1), Netherlands (1), New zealand (1), Portugal (1), Spain (1) and United states of America (1).
Pre-assignment Details: The study was planned to be conducted in 3 separate cohorts: cohort 1, 2 and 3 however, due to early termination of the study, cohort 3 was not enrolled. Participants were randomized in a 1:1 fashion to either Cohort 1 or 2. In each cohort participants were further randomized to receive either Belcesiran or placebo. Randomization was stratified based on fibrosis stage (METAVIR Score F1, F2, F3, or F4) in both cohorts 1 and 2
Groups:
- Pooled Placebo: All participants in cohort 1 and 2 received belcesiran matched placebo as subcutaneous injection, in Cohort 1 participants received monthly dosing for the first 24 weeks and then shifted to quarterly dosing thereafter until week 96 and in Cohort 2 participants received monthly dosing for the first 48 weeks and then shifted to quarterly dosing thereafter until week 96. Due to study termination participants were followed up to 2 months.
- Cohort 1: Belcesiran: Participants received a fixed dose of belcesiran 210 milligrams (mg) injection monthly for the first 24 weeks and then shifted to quarterly dosing thereafter until week 96.
- Cohort 2: Belcesiran: Participants received a fixed dose of belcesiran 210 mg injection subcutaneously monthly for the first 48 weeks and then shifted to quarterly dosing thereafter until week 96.
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Started | 5 | 5 | 6
Safety Population | 5 | 5 | 6
Completed | 0 | 0 | 0
Not Completed | 5 | 5 | 6
Not completed — Study terminated by sponsor | 2 | 2 | 5
Not completed — Withdrawal by Subject | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population is defined as all participants randomly assigned to study intervention who had received at least 1 dose of the study drug (belcesiran or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran | Total
Number analyzed (Participants) | 5 | 5 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (17.31) | 57.2 (10.18) | 52.5 (11.86) | 50.1 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
  Male | 4 | 2 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 5 | 6 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5 | 5 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: Number of TEAEs and SAEs is presented. An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs were defined as TEAEs if they had a start date on or after the administration of study drug during the treatment period, or if they occurred prior to the administration of study drug and worsened in severity/grade or relationship to the study intervention after the administration of study intervention during the treatment period. A SAE was defined as any untoward medical occurrence that, at any dose: a) resulted in death, b) is life-threatening, c) required inpatient hospitalization or prolongation of existing hospitalization, d) resulted in persistent disability/incapacity, e) was a congenital anomaly/birth defect.
Time Frame: Up to 2.6 years
Population: Safety population included all participants randomly assigned to study intervention and who received at least 1 dose of belcesiran/placebo.
Measure: Number; unit: Events
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 5 | 5 | 6
Events
  TEAE | 27 | 80 | 43
  SAE | 0 | 7 | 5

2. Primary Outcome: Number of Participants With TEAEs and SAEs
Description: Number of participants with TEAEs and SAEs is presented. An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs were defined as TEAEs if they had a start date on or after the administration of study drug during the treatment period, or if they occurred prior to the administration of study drug and worsened in severity/grade or relationship to the study intervention after the administration of study intervention during the treatment period. A SAE was defined as any untoward medical occurrence that, at any dose: a) resulted in death, b) is life-threatening, c) required inpatient hospitalization or prolongation of existing hospitalization, d) resulted in persistent disability/incapacity, e) was a congenital anomaly/birth defect.
Time Frame: Up to 2.6 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 5 | 5 | 6
Participants
  TEAE | 5 | 5 | 5
  SAE | 0 | 2 | 2

3. Primary Outcome: Change From Baseline in Pulmonary Function Tests (PFTs): Forced Vital Capacity (FVC)
Description: Change in FVC from baseline (Day 1) to week 96 is presented. FVC is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration, that is, VC performed with a maximally forced expiratory effort.
Time Frame: Baseline (Day 1), week 96
Population: Safety population included all participants randomly assigned to study intervention and who received at least 1 dose of belcesiran/placebo. Overall number of participants analyzed = Participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Liters (L) | -0.410 | -0.250 (0.0424) |

4. Primary Outcome: Change From Baseline in PFT: Forced Expiratory Volume in One Second (FEV1)
Description: Change in FEV1 from baseline (Day 1) to week 96 is presented. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
L | -0.210 | -0.290 (0.2263) |

5. Primary Outcome: Change From Baseline in PFT: FEV1/FVC Ratio
Description: Change in FEV1/FVC ratio from baseline (Day 1) to week 96 is presented. FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC is the maximal volume of air exhaled with maximally forced effort from a maximal inspiration, that is, VC performed with a maximally forced expiratory effort.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio of FEV1/FVC
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Ratio of FEV1/FVC | 0.020 | -0.055 (0.0778) |

6. Primary Outcome: Change From Baseline in PFT: Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO)
Description: Change in DLCO from baseline (Day 1) to week 96 is presented. DLCO is a measure of the quantity of carbon monoxide (CO) transferred per minute from alveolar gas to red blood cells (specifically hemoglobin) in pulmonary capillaries. It is expressed as millimoles per minute per kilopascal (mmol/min/kPa).
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/min/kPa
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
mmol/min/kPa | -1.89497 | -1.01110 (0.146774) |

7. Primary Outcome: Change From Baseline in 12 -Lead Electrochardiograms (ECGs): Mean Heart Rate
Description: Change from baseline (Day 1) to week 96 in mean heart rate is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
beats per minute | -10.0 | 1.0 |

8. Primary Outcome: Change From Baseline in 12 -Lead ECGs: Mean Ventricular Rate
Description: Change from baseline (Day 1) to week 96 in mean ventricular rate is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
beats per minute | -10.0 | 1.0 |

9. Primary Outcome: Change From Baseline in 12 -Lead ECGs: PR Interval, QRS Interval, QT Interval, QTcF Interval and RR Interval
Description: Change from baseline (Day 1) to week 96 in PR interval, QRS interval, QT interval, QTcF interval and RR interval is presented.
Time Frame: Baseline (Day 1), week 96
Population: Safety population included all participants randomly assigned to study intervention and who received at least 1 dose of belcesiran/placebo. Overall number of participants analyzed = Participants with available data for the outcome measure and number analyzed = participants with available data for each category.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
millisecond (msec)
  PR interval: number analyzed (Participants) | 1 | 0 | 0
  PR interval | -4.0 |  |
  QRS interval | 10.0 | 21.0 |
  QT interval | 26.0 | 17.0 |
  QTcF interval | -1.0 | 21.0 |
  RR interval | 224.0 | -8.0 |

10. Primary Outcome: Number of Participants With Physical Examination Findings
Description: Number of participants with physical examination findings at week 96 is presented. The data is presented under categories:a) Normal, b) Abnormal, not clinically significant, c) Abnormal, clinically significant.
Time Frame: At week 96
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Participants
  Normal | 1 | 1 | 0
  Abnormal, not clinically significant | 0 | 1 | 0
  Abnormal, clinically significant | 0 | 0 | 0

11. Primary Outcome: Change From Baseline in Vital Signs: Diastolic Blood Pressure and Systolic Blood Pressure
Description: Change from baseline (Day 1) to week 96 in diastolic blood pressure and systolic blood pressure is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
millimeters of mercury (mmHg)
  Diastolic blood pressure | 2.0 | 17.0 |
  Systolic blood pressure | 13.0 | 5.0 |

12. Primary Outcome: Change From Baseline in Vital Signs: Heart Rate
Description: Change from baseline (Day 1) to week 96 in heart rate is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
beats per minute | 1.0 | 21.0 |

13. Primary Outcome: Vital Signs: Height at Baseline
Description: Height at baseline is presented.
Time Frame: Baseline (Day 1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 5 | 5 | 6
Centimeter (cm) | 178.0 (11.07) | 167.8 (9.93) | 173.0 (13.48)

14. Primary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: Change from baseline (Day 1) to week 96 in respiratory rate is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
breaths per minute | 5.0 | 1.0 |

15. Primary Outcome: Change From Baseline in Vital Signs: Temperature
Description: Change from baseline (Day 1) to week 96 in temperature is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degree celsius
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
Degree celsius | 0.30 | -0.40 |

16. Primary Outcome: Change From Baseline in Vital Signs: Weight
Description: Change from baseline (Day 1) to week 96 in weight is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 1 | 0
kilograms (kg) | 10.70 | 0.20 |

17. Primary Outcome: Change in Clinical Laboratory Tests: Alanine Aminotransferase, Alkaline Phosphatase, Aspartate Aminotransferase, Creatine Kinase, Glutamate Dehydrogenase, Lactate Dehydrogenase, Biomarker Creatine Kinase (M30) and Biomarker Creatine Kinase (M65)
Description: Change from baseline (Day 1) to week 96 in alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, creatine kinase, glutamate dehydrogenase, lactate dehydrogenase, biomarker creatine kinase (M30) and biomarker creatine kinase (M65) is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Units per liter (U/L)
  Alanine aminotransferase | -8.0 | -10.5 (7.78) |
  Alkaline phosphatase | 26.0 | 0.0 (29.70) |
  Aspartate aminotransferase | -5.0 | -10.5 (6.36) |
  Creatine kinase | -226.0 | -3.0 (8.49) |
  Glutamate dehydrogenase | 0.0 | -4.5 (0.71) |
  Lactate dehydrogenase: number analyzed (Participants) | 0 | 2 | 0
  Lactate dehydrogenase |  | 0.5 (19.09) |
  Biomarker creatine Kinase (M30): number analyzed (Participants) | 0 | 2 | 0
  Biomarker creatine Kinase (M30) |  | -149.5 (210.01) |
  Biomarker creatine kinase (M65): number analyzed (Participants) | 0 | 2 | 0
  Biomarker creatine kinase (M65) |  | -166.180 (329.3703) |

18. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Albumin, Apolipoprotein A1, Protein, Biomarker Haptoglobin
Description: Change from baseline (Day 1) to week 96 in albumin, apolipoprotein A1, protein and biomarker haptoglobin is presented.
Time Frame: Baseline (Day 1), week 96
Population: Safety population included all participants randomly assigned to study intervention and who received at least 1 dose of belcesiran/placebo. Overall number of participants analyzed = Participants with available data for the outcome measure and number analysed = participants with avaialble data for each category.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Grams per liter (g/L)
  Albumin | -1.0 | 3.5 (0.71) |
  Apolipoprotein A1 | -0.030 | 0.180 (0.1838) |
  Protein | -2.0 | 7.5 (7.78) |
  Biomarker haptoglobin: number analyzed (Participants) | 0 | 1 | 0
  Biomarker haptoglobin |  | -0.260 |

19. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Bilirubin, Creatinine and Direct Bilirubin
Description: Change from baseline (Day 1) to week 96 in bilirubin, creatinine and direct bilirubin is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Micromoles per liter (umol/L)
  Bilirubin | 1.710 | 3.420 (0.0000) |
  Creatinine | 1.7680 | 22.5420 (19.37755) |
  Direct bilirubin | 0.000 | 0.000 (0.000) |

20. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Chloride, Cholesterol, Glucose, Potassium, Sodium, Triglycerides and Urea Nitrogen
Description: Change from baseline (Day 1) to week 96 in chloride, cholesterol, glucose, potassium, sodium, triglycerides and urea nitrogen is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Millimoles per liter (mmol/L)
  Chloride | -2.0 | -1.5 (6.36) |
  Cholesterol | -0.12950 | 0.67340 (0.842447) |
  Glucose | 0.88800 | 0.55500 (0.078489) |
  Potassium | -0.60 | 0.40 (0.283) |
  Sodium | -2.0 | -0.5 (0.71) |
  Triglycerides | -0.01130 | 0.44070 (0.399515) |
  Urea nitrogen | 0.0000 | 2.4990 (1.00975) |

21. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Gamma Glutamyl Transferase
Description: Change from baseline (Day 1) to week 96 in gamma glutamyl transferase is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
International units per liter (IU/L) | -5.0 | -30.5 (24.75) |

22. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Basophils, Eosinophils, Leucocytes, Lymphocytes, Monocytes, Neutrophils and Platelets
Description: Change from baseline (Day 1) to week 96 in basophils, eosinophils, leucocytes, lymphocytes, monocytes, neutrophils and platelets is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
10^9 cells/liter
  Basophils | -0.020 | 0.000 (0.0141) |
  Eosinophils | -0.030 | -0.020 (0.0424) |
  Leucocytes | -1.650 | -0.600 (1.1455) |
  Lymphocytes | 0.310 | -0.130 (0.0849) |
  Monocytes | -0.010 | -0.055 (0.4738) |
  Neutrophils | -1.910 | -0.380 (0.5657) |
  Platelets | -39.0 | 1.0 (16.97) |

23. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Basophils/Leucocytes
Description: Change from baseline (Day 1) to week 96 in basophils/leucocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of basophils/leucocytes
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of basophils/leucocytes | -0.10 | 0.10 (0.424) |

24. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Eosinophils/Leucocytes
Description: Change from baseline (Day 1) to week 96 in eosinophils/leucocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils/leucocytes
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of eosinophils/leucocytes | 0.20 | -0.05 (0.212) |

25. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Haematocrit
Description: Change from baseline (Day 1) to week 96 in haematocrit is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of haematocrit
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of haematocrit | 0.0 | 2.5 (2.12) |

26. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Lymphocytes/Leucocytes
Description: Change from baseline (Day 1) to week 96 in lymphocytes/leucocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes/leucocytes
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of lymphocytes/leucocytes | 17.30 | 0.85 (4.031) |

27. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Monocytes/Leucocytes
Description: Change from baseline (Day 1) to week 96 in monocytes/leucocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of monocytes/leucocytes
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of monocytes/leucocytes | 1.20 | -0.50 (6.081) |

28. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Neutrophils/Leucocytes
Description: Change from baseline (Day 1) to week 96 in neutrophils/leucocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils/leucocytes
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of neutrophils/leucocytes | -18.70 | -0.40 (1.838) |

29. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Reticulocytes/Erythrocytes
Description: Change from baseline (Day 1) to week 96 in reticulocytes/erythrocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage of reticulocytes/erythrocytes
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Percentage of reticulocytes/erythrocytes | -0.80 | 0.30 (0.141) |

30. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Erythrocyte Mean Corpuscular Haemoglobin Concentration and Haemoglobin
Description: Change from baseline (Day 1) to week 96 in erythrocyte mean corpuscular haemoglobin concentration and haemoglobin is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
g/L
  Erythrocyte mean corpuscular haemoglobin concentration | -10.0 | 0.0 (0.0) |
  Haemoglobin | -6.0 | 9.0 (4.24) |

31. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Erythrocyte Mean Corpuscular Haemoglobin
Description: Change from baseline (Day 1) to week 96 in erythrocyte mean corpuscular haemoglobin is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
picograms (pg) | -1.0 | 0.5 (0.71) |

32. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Erythrocyte Mean Corpuscular Volume
Description: Change from baseline (Day 1) to week 96 in erythrocyte mean corpuscular volume is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
femtoliter (fL) | 2.0 | 2.5 (0.71) |

33. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Erythrocytes
Description: Change from baseline (Day 1) to week 96 in erythrocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: 10^12 cells/liter
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
10^12 cells/liter | -0.10 | 0.20 (0.141) |

34. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Specific Gravity
Description: Change from baseline (Day 1) to week 96 in specific gravity is reported.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Ratio | -0.0050 | 0.0025 (0.01061) |

35. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Urine Erythrocytes and Urine Leucocytes
Description: Change from baseline (Day 1) to week 96 in urine erythrocytes and urine leucocytes is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per high power field (/HPF)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 0 | 1 | 0
per high power field (/HPF)
  Urine erythrocytes |  | 3.0 |
  Urine leucocytes |  | 0.0 |

36. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Potential of Hydrogen (pH)
Description: Change from baseline (Day 1) to week 96 in pH is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
pH | 0.00 | -0.75 (1.061) |

37. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Activated Partial Thromboplastin Time and Prothrombin Time
Description: Change from baseline (Day 1) to week 96 in activated partial thromboplastin time and prothrombin time is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: seconds (sec)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
seconds (sec)
  Activated partial thromboplastin time | 0.40 | 1.55 (2.333) |
  Prothrombin time | -0.50 | 0.40 (0.990) |

38. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Prothrombin International Normalized Ratio
Description: Change from baseline (Day 1) to week 96 in prothrombin international normalized ratio is presented.
Time Frame: Baseline (Day 1), week 96
Population: Safety population included all participants randomly assigned to study intervention and who received at least 1 dose of belcesiran/placebo. Overall number of participants analyzed= Participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
Ratio | 0.00 | 0.00 (0.141) |

39. Primary Outcome: Change in Clinical Laboratory Tests: Alpha Fetoprotein, Biomarker Hyaluronic Acid, Biomarker Matrix Metalloproteinase 9, Biomarker Procollagen 3 N-Terminal Propeptide, Biomarker Tissue Inhibitor of Metalloproteinase 1, Complement C3a and Complement C5a
Description: Change from baseline (Day 1) to week 96 in alpha fetoprotein, biomarker hyaluronic acid, biomarker matrix metalloproteinase 9, biomarker procollagen 3 N-Terminal propeptide, biomarker tissue inhibitor of metalloproteinase 1, complement C3a and complement C5a is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanograms per milliter (ng/mL)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
nanograms per milliter (ng/mL)
  Alpha fetoprotein | 0.30 | 2.90 (2.687) |
  Biomarker hyaluronic acid: number analyzed (Participants) | 0 | 2 | 0
  Biomarker hyaluronic acid |  | 137.305 (310.3704) |
  Biomarker matrix metalloproteinase 9: number analyzed (Participants) | 0 | 2 | 0
  Biomarker matrix metalloproteinase 9 |  | -193.65 (239.356) |
  Biomarker procollagen 3 N-terminal propeptide: number analyzed (Participants) | 0 | 2 | 0
  Biomarker procollagen 3 N-terminal propeptide |  | -0.655 (0.5020) |
  Biomarker tissue inhibitor of metalloproteinase 1: number analyzed (Participants) | 0 | 2 | 0
  Biomarker tissue inhibitor of metalloproteinase 1 |  | -83.25 (8.980) |
  Complement C3a | 139.70 | -5.60 (5.657) |
  Complement C5a | 1.890 | -1.785 (0.6152) |

40. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: C-Reactive Protein
Description: Change from baseline (Day 1) to week 96 in C-reactive protein is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
mg/L | 4.30 | -0.30 (0.849) |

41. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Complement Bb
Description: Change from baseline (Day 1) to week 96 in complement Bb is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microgram per milliliter (ug/mL)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
microgram per milliliter (ug/mL) | 0.240 | 0.325 (0.2616) |

42. Primary Outcome: Change From Baseline in Clinical Laboratory Tests: Complement Total (CH50)
Description: Change from baseline (Day 1) to week 96 in CH50 is presented.
Time Frame: Baseline (Day 1), week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: equivalent unit per milliliter (U Eq/mL)
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 2 | 0
equivalent unit per milliliter (U Eq/mL) | 6.530 | -46.900 (40.1071) |

43. Primary Outcome: Cohort 1: Change From Baseline in Serum Alpha-1 Antitrypsin (AAT) Protein Concentrations
Description: Change from baseline (Day 1) to week 24 in serum AAT protein concentrations in Cohort 1 is presented.
Time Frame: Baseline (Day 1), week 24
Population: Pharmacodynamic (PD) population included all participants randomly assigned to study intervention who received at least 1 dose of belcesiran (or placebo) and at least 1 postdose PD assessment. Overall number of participants analyzed = Participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 1: Belcesiran
Number analyzed (Participants) | 4
g/L | -0.30 (0.120)

44. Primary Outcome: Cohort 2: Change From Baseline in Serum AAT Protein Concentrations
Description: Change from baseline (Day 1) to week 48 in serum AAT protein concentrations in Cohort 2 is presented.
Time Frame: Baseline (Day 1), week 48
Population: PD population included all participants randomly assigned to study intervention who received at least 1 dose of belcesiran (or placebo) and at least 1 postdose PD assessment. Overall number of participants analyzed = Participants with available data for the outcome measure.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Cohort 2: Belcesiran
Number analyzed (Participants) | 3
g/L | -0.50 (0.094)

45. Secondary Outcome: Change From Baseline in Liver Fibrosis Ishak Score
Description: Change from Baseline up until week 48 in liver fibrosis based on Ishak score is presented. The Ishak staging system for liver fibrosis is a 1995 update to the algorithm initially developed by De Groote et al. Ishak scores range from 0 (no fibrosis) to 6 (cirrhosis) which are as follows: 0-no fibrosis, 1-fibrous expansion of some portal areas, with or without short fibrous septa, 2-Fibrous expansion of most portal areas, with or without short fibrous septa, 3-Fibrous expansion of most portal areas with occasional portal-to-portal bridging, 4-Fibrous expansion of portal areas with marked bridging (portal to portal as well as portal to central), 5-Marked bridging (portal-portal and/or portal-central) with occasional nodules (incomplete cirrhosis), 6-Cirrhosis, probable or definite.
Time Frame: Baseline (Day 1), week 48
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: unit on a score
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
Number analyzed (Participants) | 1 | 0 | 3
unit on a score | 1.0 |  | -1.0 (0.00)

ADVERSE EVENTS:
Time Frame: Up to 2.6 years
Description: Results are based on safety population. Safety Population was defined as all participants randomly assigned to study intervention and who received at least 1 dose of study drug. Presented AEs are TEAEs. AEs were defined as TEAEs if they had start date on or after administration of study drug during treatment period, or if they occurred prior to administration of study drug and worsened in severity/grade or relationship to study drug after administration during treatment period.
Arm/Group | Pooled Placebo | Cohort 1: Belcesiran | Cohort 2: Belcesiran
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 2/5 | 2/6
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=5) | Cohort 1: Belcesiran (N=5) | Cohort 2: Belcesiran (N=6)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary function test decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pooled Placebo (N=5) | Cohort 1: Belcesiran (N=5) | Cohort 2: Belcesiran (N=6)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 1 (1) | 2 (2) | 0 (0)
Hyaluronic acid increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Pulmonary function test decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Complement factor C4 increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Enzyme level increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Faecal volume increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lung diffusion test decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Serum procollagen type III N-terminal propeptide increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Alpha-2 macroglobulin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site discoloration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (5)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1)
Varices esophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04764448/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/48/NCT04764448/SAP_001.pdf